CLINICAL TRIAL: NCT04634903
Title: Comparing Two Online Single-Session Interventions for Adolescent Depression: Outcomes of a Randomized Trial
Brief Title: Testing Scalable, Single-Session Interventions for Adolescent Depression in the Context of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: University of Denver (Other)
Responsible Party: Principal Investigator, Jessica Schleider, Assistant Professor of Psychology, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1505797-3
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Depression
Keywords: single-session interventions
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the Behavioral Activation SSI (BA-SSI), Growth Mindset SSI (GM-SSI), or the Supportive Therapy SSI (ST-SSI; each 30 minutes in length).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supportive Therapy SSI (ST-SSI) (Active Comparator): The web-based supportive therapy (ST-SSI) intervention, called the Sharing Feelings Intervention, is designed to mimic supportive therapy (ST). The goals of the ST intervention are to encourage participants to identify and express feelings to close others; the intervention does not teach or emphasize specific skills or beliefs. In previous clinical trials, ST has resulted in significantly fewer reductions in youth internalizing problems compared to cognitive-behavioral and growth mindset interventions. The ST-SSI is designed to control for nonspecific aspects of intervention, including engagement in a computer program. It includes the same number of reading and writing activities as the other SSIs.
  Interventions: Behavioral: Supportive Therapy SSI
- Behavioral Activation SSI (BA-SSI) (Experimental): The BA-SSI include 5 elements: (1) An introduction to the program's rationale: that engaging in value-based activities can combat sad mood and low self-esteem; (2) Psychoeducation about depression, including how behavior shapes feelings and thoughts; (3) A life values assessment, where youth identify key areas from which they draw enjoyment and meaning; (4) Creation of an activity hierarchy, where youth identify and personalize (in guided exercises) 3 activities to target for change; and (5) An exercise in which youths write about benefits that might result from engaging in each activity; an obstacle that might keep them from doing the activities; and a strategy for overcoming identified obstacles.
  Interventions: Behavioral: Behavioral Activation SSI
- Growth Mindset SSI (GM-SSI) (Experimental): Program includes: An introduction to the brain and a lesson on neuroplasticity; Testimonials from older youths who describe their views that traits are malleable Further stories by older youths, describing times when they used "growth mindsets" to persevere during social/emotional setbacks; Study summaries noting how/why personality can change; And an exercise in which youths write notes to younger students, using scientific information to explain people's capacity for change.
  Interventions: Behavioral: Growth Mindset SSI

INTERVENTIONS:
Behavioral: Supportive Therapy SSI — Online, 30-minute self-administered program for youth
  Other Names: Sharing Feelings SSI; ST-SSI
  Arms: Supportive Therapy SSI (ST-SSI)
Behavioral: Behavioral Activation SSI — Online, 30-minute self-administered program for youth
  Other Names: Activate Action; BA-SSI
  Arms: Behavioral Activation SSI (BA-SSI)
Behavioral: Growth Mindset SSI — Online, 30-minute self-administered program for youth
  Other Names: Project Personality; GM-SSI
  Arms: Growth Mindset SSI (GM-SSI)

SUMMARY:
Most mental health problems emerge by age 14, often leading to chronic impairments and adverse impacts for individuals, families, and societies. Any action-focused path to reducing the need-to-access gap will require moving beyond the dominant settings, formats, and systems that have constrained intervention delivery to date. In a fully-online trial, youths ages 13-16 will be randomized to 1 of 3 self-administered single-session interventions (SSIs): a behavioral activation SSI, targeting behavioral MD symptoms; an SSI teaching growth mindset, targeting cognitive MD symptoms; or a control SSI. The investigators will test each SSI's relative benefits, versus the control, on depressive symptoms and proximal outcomes such as hopelessness. Results will reveal whether SSIs that were designed to address behavioral versus cognitive symptoms differentially benefit adolescents with elevated depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* are fluent in English
* have consistent internet and computer/laptop/smartphone access
* report elevated depressive symptoms (a score of >2 on the Patient Health Questionnaire-2 item version [PHQ-2])

Exclusion Criteria:

* fail to meet the above-listed inclusion criteria
* exit the study prior to condition randomization
* respond with either copy/pasted responses from text earlier in the intervention to any of free response questions
* obvious lack of English fluency in open response questions
* responding with random text in open response questions
* duplicate responses from the same individual in baseline or follow-up surveys

We will also exclude for primary analyses (but may run sensitivity analyses including them) any participants who provide responses of fewer than 3 words to writing prompts that ask for at least 2 sentences or more.

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2452 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Schleider, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Protocol and statistical plan have been posted to Open Science Framework prior to the start of this trial as part of study pre-registration (https://osf.io/kumdv/). Code will be made available upon publication of trial results.
URL: https://osf.io/8mk6x

REFERENCES:
- [Derived] Szkody E, Chang YW, Schleider JL. Serving the Underserved? Uptake, Effectiveness, and Acceptability of Digital SSIs for Rural American Adolescents. J Clin Child Adolesc Psychol. 2025 Sep-Oct;54(5):541-554. doi: 10.1080/15374416.2023.2272935. Epub 2023 Nov 6. PMID 37931065
- [Derived] Ahuvia IL, Mullarkey MC, Sung JY, Fox KR, Schleider JL. Evaluating a treatment selection approach for online single-session interventions for adolescent depression. J Child Psychol Psychiatry. 2023 Dec;64(12):1679-1688. doi: 10.1111/jcpp.13822. Epub 2023 May 14. PMID 37183368
- [Derived] Cohen KA, Shroff A, Nook EC, Schleider JL. Linguistic distancing predicts response to a digital single-session intervention for adolescent depression. Behav Res Ther. 2022 Dec;159:104220. doi: 10.1016/j.brat.2022.104220. Epub 2022 Oct 20. PMID 36323056
- [Derived] Schleider JL, Mullarkey MC, Fox KR, Dobias ML, Shroff A, Hart EA, Roulston CA. A randomized trial of online single-session interventions for adolescent depression during COVID-19. Nat Hum Behav. 2022 Feb;6(2):258-268. doi: 10.1038/s41562-021-01235-0. Epub 2021 Dec 9. PMID 34887544

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Therapy SSI (ST-SSI) | Behavioral Activation SSI (BA-SSI) | Growth Mindset SSI (GM-SSI)
Started | 818 | 821 | 813
Completed | 669 | 732 | 653
Not Completed | 149 | 89 | 160

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supportive Therapy SSI (ST-SSI) | Behavioral Activation SSI (BA-SSI) | Growth Mindset SSI (GM-SSI) | Total
Number analyzed (Participants) | 818 | 821 | 813 | 2452
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 818 | 821 | 813 | 2452
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 723 | 718 | 719 | 2160
  Male | 87 | 86 | 78 | 251
  Other | 2 | 12 | 7 | 21
  Prefer not to say | 6 | 5 | 9 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Category options were not mutually exclusive; respondents could select multiple races/ethnicities.
  Participants
    American Indian/Alaska Native | 36 | 27 | 29 | 92
    Asian | 101 | 109 | 100 | 310
    Hispanic | 159 | 164 | 148 | 471
    Native Hawaiian/Pacific Islander | 14 | 11 | 14 | 39
    White | 546 | 536 | 550 | 1632
    Black | 85 | 84 | 88 | 257
    Other | 19 | 17 | 11 | 47
    Prefer not to say | 9 | 5 | 10 | 24
Region of Enrollment [Number; unit: participants]
  United States | 818 | 821 | 813 | 2452

OUTCOME MEASURES:

1. Primary Outcome: Change in Adolescent Depressive Symptom Severity
Description: The Children's Depression Inventory (CDI) 2 - short form (CDI-SF) is a reliable, valid measure of youth depression severity, normed for youth age and sex and yielding raw scores ranging from 0-24, where higher scores indicate more severe symptoms of depression.
Time Frame: Pre-SSI to 3-month follow-up
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Supportive Therapy SSI (ST-SSI) | Behavioral Activation SSI (BA-SSI) | Growth Mindset SSI (GM-SSI)
Number analyzed (Participants) | 818 | 821 | 813
Score on a scale
  Pre-Intervention CDI-II Score | 14.31 (4.12) | 14.15 (4.06) | 14.22 (4.13)
  3-month follow up CDI-II score | 12.57 (4.97) | 11.47 (5.04) | 11.58 (5.08)

2. Secondary Outcome: Change in State Hope Scale - Pathways Subscale
Description: The State Hope Scale - Pathways Subscale asks participants to rate 3 statements based on how they think about themselves right now. Participants rate the 3 statements on an 8 point scale ranging from 0 (Definitely False) to 7 (Definitely True). Total score ranges, reflecting the average across all items, range from 0-7, with higher scores representing more flexible/greater perceived pathways to solving one's problems.
Time Frame: Pre-SSI to Immediately Post-SSI; Pre-SSI to 3-month follow-up
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Supportive Therapy SSI (ST-SSI) | Behavioral Activation SSI (BA-SSI) | Growth Mindset SSI (GM-SSI)
Number analyzed (Participants) | 818 | 821 | 813
Score on a scale
  Pre-intervention | 3.88 (1.39) | 3.93 (1.40) | 3.96 (1.44)
  Post-intervention | 5.26 (1.52) | 5.68 (1.43) | 5.50 (1.48)
  3-month follow up | 4.89 (1.64) | 5.06 (1.63) | 5.17 (1.65)

3. Secondary Outcome: Change in Beck Hopelessness Scale - 4 Item Version
Description: 4 item version (BHS-4; referenced as 'How I Think Scale' in appended materials): This scale asks participants to rate 4 statements based on their sense of hopelessness. Participants rate the 4 statements on a 4 point scale ranging from 0 (Absolutely Disagree) to 3 (Absolutely Agree). Average scores across all items range from 0 to 3, with a higher score indicating greater levels of hopelessness.
Time Frame: Pre-SSI to Immediately Post-SSI; Pre-SSI to 3-month follow-up
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Supportive Therapy SSI (ST-SSI) | Behavioral Activation SSI (BA-SSI) | Growth Mindset SSI (GM-SSI)
Number analyzed (Participants) | 818 | 821 | 813
Score on a scale
  Pre-intervention | 1.71 (0.76) | 1.72 (0.77) | 1.72 (0.76)
  Post-intervention | 1.36 (0.75) | 1.22 (0.73) | 1.21 (0.72)
  3-month follow up | 1.51 (0.82) | 1.37 (0.80) | 1.39 (0.83)

4. Secondary Outcome: Program Feedback Scale
Description: The PFS asks youth to rate agreement with 7 statements indicating perceived acceptability of an SSI (e.g. "I enjoyed the program") on a 5-point Likert scale (1="really disagree"; 5="totally agree"). A score of 3.5/5 or above on any given PFS item is interpreted as an "acceptable" rating on that item. Scores are calculated at the item-level, and higher scores reflect greater acceptability for each item.
Time Frame: Immediately Post-SSI only
Population: Mean item-level scores ranging from 1-5 are reported for each of 7 PFS items. Items were administered at post-intervention only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Therapy SSI (ST-SSI) | Behavioral Activation SSI (BA-SSI) | Growth Mindset SSI (GM-SSI)
Number analyzed (Participants) | 630 | 729 | 653
score on a scale
  PFS Item 1: Enjoyed Program | 3.80 (0.79) | 3.93 (0.73) | 3.83 (0.77)
  PFS item 2: Understood Program | 4.54 (0.56) | 4.46 (0.49) | 4.48 (0.64)
  PFS Item 3: Program was Easy to Use | 4.46 (0.64) | 4.42 (0.59) | 4.48 (0.64)
  PFS Item 4: I tried my hardest on the program | 4.45 (0.65) | 4.42 (0.69) | 4.45 (0.67)
  PFS item 6: I would recommend this program to a friend | 3.97 (0.95) | 4.12 (0.89) | 3.93 (1.00)
  PFS item 5: This program would be helpful to other kids | 4.24 (0.81) | 4.30 (0.76) | 4.20 (0.83)
  PFS item 7: I agree with the program's message | 4.50 (0.62) | 4.54 (0.57) | 4.47 (0.70)

5. Other Pre Specified Outcome: Change in Behavioral Activation for Depression Scale - Short Form
Description: Youths' approach versus disengagement from rewarding activities will be assessed via the BADS-SF, a 9-item self-report questionnaire with strong reliability, predictive validity, and sensitivity to change following BA for adolescent depression symptoms. The BADS-SF has two subscales, both of relevance to this study: Activation (goal-directed engagement in rewarding activities) and Avoidance (engagement in rumination and avoidance rather than active coping).
Time Frame: Pre-SSI to 3-month follow-up
Reporting Status: Not Posted, anticipated posting 2021-09

6. Other Pre Specified Outcome: Change in Self-Injurious Thoughts and Behaviors Interview-Short Form (SITBI-SF)
Description: Four items from a self-report version of the SITBI-SF were used to assess lifetime history of suicide ideation, suicide attempts, and deliberate self-harm. The SITBI-SF is a widely used measure of the continuum of suicidality and self-harm and has demonstrated high test-retest reliability, high internal consistency, and moderate-to-high concurrent validity. Score range for this measure can range widely (per wide variation in instances of self-harming behaviors across one's lifetime); thus, we anticipate a minimum score of 0 and are unable to predict the top (maximum) score.
Time Frame: Pre-SSI to 3-month follow-up
Reporting Status: Not Posted, anticipated posting 2021-12

7. Other Pre Specified Outcome: Change in Implicit Personality Theory Questionnaire
Description: The IPTQ asks youth to rate the extent of their agreement with three statements linked to the malleability of personality, using a 1-to-7 Likert scale (e.g. "Your personality is something about you that you can't change very much.") Higher mean scores (range: 1-7) on these three items indicate a stronger fixed personality mindset, lower scores, a stronger growth personality mindset.
Time Frame: Pre-SSI, Immediately Post-SSI
Reporting Status: Not Posted, anticipated posting 2021-09

8. Other Pre Specified Outcome: Demographic Questions
Description: Participants will be asked to report demographic information including age, sex assigned at birth, gender identity, primary language, school grade, race/ethnicity, sexual/romantic attraction, experiences, and orientation, and zip code. This measure will also assess mental health treatment history and pubertal status.
Time Frame: Pre-SSI only
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Perceived Socioeconomic and Social Status
Description: Immediately pre-intervention, participants will be asked to rate their perceived socioeconomic and social status using the two items from the MacArthur Scale of Subjective Social Status-Youth Version. Respondents indicate where they see themselves on a ladder with 10 rungs (range: 1 to 10 for both items, where 1 = families with most money/education/jobs and youth with highest respect/grades/social standing; 10 = families with least money/education/jobs and youth with lowest respect/grades/social standing).
Time Frame: Pre-SSI only
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Multidimensional Peer Victimization Scale
Description: The MVPS is a self-report scale assessing adolescents' experiences of peer victimization. This study will include the social manipulation, verbal victimization, and physical victimization scales, totaling 12 items (4 items per subscale). Higher scores on any given subscale indicate more frequent victimization of specific type. Adolescents rate how often peers have victimized them in various ways in the past year (e.g. "called me names"; "tried to turn my friends against me").
Time Frame: Pre-SSI only
Reporting Status: Not Posted

11. Other Pre Specified Outcome: UCLA Loneliness Scale
Description: The ULS is a widely used self-report scale of loneliness in adolescents. The brief 8-item version will be used here. Adolescents rate agreement with 8 items reflecting loneliness (e.g. "I feel left out"; "I feel isolated from others"). Higher summed-scores across all 8 items reflect higher levels of loneliness. The ULS has shown adequate reliability and validity in adolescent samples.
Time Frame: Pre-SSI only
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Self-Referential Encoding Task (SRET)
Description: The SRET is a web-based behavioral measure of self-referent information processing biases that assesses judgements of self-descriptiveness, response latencies and free recall of emotionally valanced stimuli. Participants make decisions about whether positive and negative adjectives are self-descriptive. Participants view various adjectives (26 positive adjectives, 26 negative adjectives) one at a time and make rapid judgments about whether or not each word presented described themselves following word offset. Participants will be told to use the Q or P keys on their keyboard to answer whether the word described them or not. Each trial will be followed by a 1,500 ms intertrial interval.
Time Frame: Pre-SSI
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Discrimination
Description: The Expanded Everyday Discrimination Scale will be measured pre-intervention to gauge the levels of relatively minor, every-day, chronic discrimination experienced by participants. The original scale (Williams et al., 1997) asks participants, "In your day-to-day life, how often do any of the following things happen to you?" for 9 items (e.g. "you are treated with less courtesy than other people are") on a 5-point Likert scale (1= "never"; 6 = "almost every day"). These items assess the participant's observations about how others treat and act around them on a daily basis. The expanded version of this scale includes a 10th item, "You are followed around in stores." Scores on the Expanded Everyday Discrimination Scale range from 10-60, with higher scores indicating higher levels of chronic discrimination experienced by participants. Respondents are also asked to identify what they believe to be the main reason(s) for these experiences (e.g. gender, race, age, etc.).
Time Frame: Pre-SSI
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Generalized Anxiety Disorder 7 (GAD-7)
Description: The GAD-7 measures the severity of clinical anxiety symptoms, based on diagnostic criteria for generalized anxiety disorder. The GAD-7 includes 7 items asking respondents how often, during the last 2 weeks, they were bothered by each of 7 anxiety symptoms. Response options are "not at all," "several days," "more than half the days," and "nearly every day," scored as 0, 1, 2, and 3, respectively; thus total sum-scores may range from 0-21 and average scores from 0 to 3.
Time Frame: Pre-SSI
Reporting Status: Not Posted

15. Other Pre Specified Outcome: COVID-19-related Stressors
Description: Youths will self-report perceived family social status related to the COVID-19 pandemic began (ie current perceived family social status), along with which among several COVID-19-related challenges they have faced (e.g., parent has lost job; school has closed; less contact with friends; know someone who was sick with COVID-19; more conflict at home; feel bored/restless; other [free response]). Item choices will be adapted from those included in the CDC's publicly-available item bank for research on COVID-19.
Time Frame: Pre-SSI only
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in COVID-19-related Trauma Symptoms
Description: The Child Trauma Screen-Reaction Scale (CTS-RS) is a reliable, valid self-report measure of youth traumatic stress symptom severity, including event-related somatic symptoms, intrusive memories, avoidance, sleep problems, and mood and behavioral changes. For this study, instructions will read: "For many kids and teens, the COVID-19 (or 'coronavirus') pandemic has been scary or very upsetting. Sometimes, events that are scary or upsetting can affect how people think, feel, and act. The next questions ask how you have been feeling and thinking recently." Youth will rate 6 statements describing traumatic stress symptoms (e.g., 'strong feelings in your body when you think about COVID-19 (sweating, heart beats fast, feel sick)') according to their frequency over the past 30 days (Never/Rarely; 1-2 times in the past month; 1-2 times in the past week; 3+ times per week).
Time Frame: Pre-SSI to 3-month follow-up
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Disordered Eating
Description: Disordered eating behaviors will be measured at pre-intervention and 3-month follow-up using The Dietary Restriction Screener. The DRS-2 is a 9-item measure evaluating restrictive eating, bingeing, and purging behaviors in participants. 6 items ask participants whether or not they have engaged in restrictive eating, bingeing, or purging behaviors in the past year or in the past 3 months (0 = no; 1 = yes). The other 3 items assess the frequency of these behaviors over the past 28 days.
Time Frame: Pre-SSI to 3-month follow-up
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Adverse Childhood Experiences (ACEs) Scale
Description: The ACEs questionnaire asks about exposure to violence, childhood emotional, physical, or sexual abuse, and household dysfunction during childhood. ACEs have shown robust associations with a range of adverse health and behavioral outcomes across the lifespan [yes/no]. Questions asked in this measure include:
  At any point since you were born…
  1. Did you often or very often feel that… No one in your family loved you or thought you were important or special? or Your family didn't look out for each other, feel close to each other, or support each other?
  2. Were your parents ever separated or divorced?
  3. Did you live with anyone who was a problem drinker or alcoholic, or who used street drugs?
  4. Was a household member depressed or mentally ill, or did a household member attempt suicide?
  5. Did a household member go to prison?
Time Frame: Pre-SSI only
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Brief Screener for Tobacco, Alcohol, and Other Drugs (BSTAD)
Description: The BSTAD questionnaire asks respondents to report retrospectively on their personal and friends' tobacco and drug use over the past year the past year (yes/no), including questions about how frequently (in days) the respondent recalls using alcohol, tobacco, and other drugs.
Time Frame: Pre-SSI only
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Perceived Pre-to-post SSI Change Items
Description: Participants rate their perceived changes in levels of pre- to post-SSI hopelessness and ability to solve problems. The questions are:
  Compared to before doing this activity, to what extent are you feeling hopeless right now? (Response options: much more hopeless = -2; a little more hopeless = -1; the same amount of hopeless = 0; a little less hopeless = 1; a lot less hopeless = 2).
  Compared to before doing this activity, to what extent are you able to solve the problems facing you right now? (Response options: Much less able to solve problems = -2; a little less able to solve problems = -1; the same amount able to solve problems = 0; a little more able to solve problems = 1; a lot more able to solve problems = 2)
Time Frame: Immediately Post-SSI only
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months (baseline through final follow up in the trial)
Arm/Group | Supportive Therapy SSI (ST-SSI) | Behavioral Activation SSI (BA-SSI) | Growth Mindset SSI (GM-SSI)
All-Cause Mortality (participants affected / at risk) | 0/818 | 0/821 | 0/813
Serious Adverse Events (participants affected / at risk) | 0/818 | 0/821 | 0/813
Other Adverse Events (participants affected / at risk) | 0/818 | 0/821 | 0/813

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT04634903/Prot_SAP_000.pdf